CLINICAL TRIAL: NCT05629221
Title: Organisational Models Supported by Technology for the Management of Diabetic Disease and Its Complications in a Diabetic Clinic Setting. A Randomised Controlled Trial Targeting Type 2 Diabetes Individuals With Non-ideal Glycemic Values
Acronym: Telemechron
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other)
Collaborators: Fondazione Bruno Kessler (Other); Provincia Autonoma di Trento (Other Government); TrentinoSalute4.0 (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Inchiostro Sandro, Doctor, Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Telemechron - A765; NET-2018-12367206 - WP4 (Other: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento)
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Diabetes type2
Keywords: telemedicine; smartphone; mHealth; mobile applications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TreC Diabete App users (Experimental): Sixty individuals allocated to the intervention group are prescribed with the TreC Diabete App for 12 months, one of the App created within the so-called TreC platform, which enables citizens from PAT to access, manage and share information about their health and wellbeing in the context of telemedicine. The use of the App is additional to the standard care, based on the integrated preventive and diagnostic care pathway (called "Percorsi Preventivi Diagnostici Terapeutici Assistenziali - PPDTA" in Italian).An appointment with the outpatient diabetes clinic staff is scheduled at 6 and 12 month from the first visit (taking place within 30 days of the study entry), either through telemedicine (remote visit) or face-to-face.
  Interventions: Other: TreC Diabete App
- non-App users (No Intervention): Sixty individuals are allocated to the control group. These participants will receive standard care, which is the best care for T2DM in line with the integrated preventive and diagnostic care pathway (called "Percorsi Preventivi Diagnostici Terapeutici Assistenziali - PPDTA" in Italian).An appointment with the outpatient diabetes clinic staff is scheduled at 6 and 12 month from the first visit (taking place within 30 days of the study entry), either through telemedicine (remote visit) or face-to-face. Participants are asked to register their data as per routine (e.g. paper diary).

INTERVENTIONS:
Other: TreC Diabete App — Participants can download the App from Google Play or Apple Store and activate the App as soon as the clinician provides them a unique activation code, created through an online medical dashboard. The dashboard allows the interaction between healthcare staff and the participant through the use of a chat or a video-chat. Participants are asked to register some information in the App at set times (e.g. blood pressure). Reminders are periodically sent to remember the participants to perform some tasks. Clinicians will periodically check the information entered by the participant (min frequency 45 days).
  Arms: TreC Diabete App users

SUMMARY:
The goal of this randomised trial is to evaluate the impact of using a digital platform called "TreC Diabete" embedded into a novel organizational asset for poorly controlled type 2 diabetes individuals in the Autonomous Province of Trento (PAT). The main question aims to answer whether individuals using the "TreC Diabete" platform will improve their haemoglobin glycated level (Hb1Ac) at 12-month post-randomisation. Participants will be asked to perform some tasks and to share their data with the healthcare staff members through the platform. Control group will receive standard care.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a non-communicable disease representing one of the most serious public health challenges of the 21st century. Its incidence continues to rise in both developed and developing countries, causing the death of 1.5 million people every year. The use of technology (e.g. Smartphone application - App) in the health field has progressively increased as it has been proved effective in helping some individuals manage their long-term diseases. Therefore, it has the potential to reduce health service utilization and its related costs. The objective of this study is to evaluate the impact of using a digital platform called "TreC Diabete" embedded into a novel organizational asset targeting poorly controlled T2DM individuals in the Autonomous Province of Trento (PAT), Italy.This trial was designed as a multi-center, open-label, randomised, superiority study with two parallel-groups and a 1:1 allocation ratio. Individuals regularly attending outpatients diabetes clinics, providing informed consent are randomised to be prescribed TreC Diabete platform or not as part of their personalised care plan. Healthcare staff members will remotely assess the data shared by the participants through the App by using a dedicated online medical dashboard. The primary end-point is the evaluation of the Hb1Ac level at 12-month post-randomisation. Data will be analysed on an intention-to-treat (ITT) basis.This trial is the first conducted in the PAT for the use of an App specifically designed for individuals with poorly controlled T2DM. If the effects of introducing this specific App within a new organizational asset are positive, the digital platform will represent a possible way for people diagnosed with T2DM to better manage their health in the future. Results will be disseminated through conferences and peer-reviewed journals once the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with T2DM;
* aged ≥ 18 and ≤ 85 years old;
* having an HbA1c level >7% (53 mmol/mol) and <12% (108 mmol/mol);
* being able to walk without walking aids;
* having provided written informed consent;
* having a smartphone or a tablet and being able to download the App that will be used to insert the required data.

Exclusion Criteria:

* having a BMI <18 Kg/m² and >45 Kg/m²;
* having a sBP <100 or >200 mmHg and/or dBP <50 or >120 mmHg;
* being diagnosed with a stage 5 CKD*
* being diagnosed with a NYHA stage IV;
* poor collaboration (ie unwilling to modify the actual plan of control and therapy, even if not ideal) for which adherence to the study is unlikely
* having no possibility of using a smartphone or a tablet
* having medical conditions affecting the study participation (i.e. life expectancy < 1 year)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin glycated (Hb1Ac) mean changes | 12 months
  Difference in the participants' HbA1c level between the two arms. Blood test carried out by qualified nurses and processes by the local analysis laboratory. Blood tests results are automatically registered on the Hospital Information System (HIS) and reviewed by clinicians and research staff involved in the study.

SECONDARY OUTCOMES:
Proportion of participants with Hb1Ac <53mmol/mol | 12 months
  Proportion of participants with Hb1Ac <53mmol/mol within the two arms
Hb1Ac mean changes | 3 months, 6 months and 9 months
  Difference in the participants' HbA1c level at different time frame other than at 12 months
Number of hypoglycemic episodes | 12 months
  Frequency of hypoglycemic episodes within the two arms
Number of subjects reaching targeted lipid profile | 12 months
  Proportion of participants reaching the targeted lipid profile (LDL level <70 mg/dl and non-HDL cholesterol level <100 mg/dl)
Number of subjects reaching targeted blood pressure levels | 3 months, 6 months, 9 months, 12 months
  Proportion of participants reaching the targeted BP levels (sBP <130mmHg or <140 if ≥65 years old) and dBP <80mmHg)
Effect on weight | 3 months, 6 months, 9 months and 12 months
  Effect on weight for the app users
Level of physical activity | 3 months, 6 months, 9 months and 12 months
  Information collected through specific questionnaires
Quality of life score changes | 12 months
  Changes in quality of life scores for participants of both arms through a specific questionnaire
Satisfaction and usability score of the App | 12 months
  Satisfaction and usability score of the App in the intervention group only
Number of telemedicine visits between participants and nurses/clinicians and chat interactions | 3 months, 6 months, 9 months and 12 months
  Process indicator outcome
Number of (tele)specialist consultations | 3 months, 6 months, 9 months and 12 months
  Process indicator outcome
Number of changes in the therapeutic plan | 3 months, 6 months, 9 months and 12 months
  Process indicator outcome: number of changes in the therapeutic plan (e.g. drug prescription and dosage)
Time spent for telemedicine visits | 6 months
  Process indicator outcome: amount of time spent for telemedicine visits (calculated on the basis of the average time spent to deliver eight consecutive nursing visits and eight consecutive medical visits)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Inchiostro, Principal Investigator — Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento
Locations (1):
- Azienda Provinciale per i Servizi Sanitari, Trento, Trentino-Alto Adige, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will not be available on an individual level. We plan to share data on their aggregated form

REFERENCES:
- [Derived] Giovanazzi A, Gios L, Mastellaro M, Gentilini MA, Valent F, Condini S, Bincoletto G, Bacchiega A, Zorzi A, Malfatti G, Perini F, Eccher C, Marchesoni M, Dall'Alda M, Orrasch M, Conforti D, Inchiostro S. Organisational models supported by technology for the management of diabetic disease and its complications in a diabetic clinic setting: study protocol for a randomised controlled trial targeting type 2 diabetes individuals with non-ideal glycaemic values (Telemechron study). Trials. 2023 Aug 10;24(1):513. doi: 10.1186/s13063-023-07515-6. PMID 37563665